CLINICAL TRIAL: NCT01942187
Title: A Comparison of Medication Augmentation and Problem Solving Therapy
Brief Title: A Comparison of Medication Augmentation and PST in the Treatment of Depression in Older Adults
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Bret Rutherford, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #6627
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Major Depressive Disorder; Dysthymic Disorder; Depressive Disorder Not Otherwise Specified (NOS)
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder | interventions — Aripiprazole; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medication Augmentation (Active Comparator): Medication augmentation with aripiprazole (Abilify) starting at 5mg/day, and increasing weekly in 5mg increments to a maximum of 15mg (10mg/day is the target dose). Under conditions of nonresponse after 6 weeks, aripiprazole will be switched for bupropion (Wellbutrin), starting at 150mg, and possibly increasing to 300mg after 2 weeks.
  Interventions: Drug: Aripiprazole; Drug: Bupropion
- Problem Solving Therapy (Active Comparator): Treatment for 12 weeks with weekly sessions of Problem Solving Therapy, with a trained therapist.
  Interventions: Behavioral: Problem Solving Therapy

INTERVENTIONS:
Drug: Aripiprazole — Medication augmentation with Abilify (aripiprazole), in participants who have not responded to Selective Serotonin Reuptake Inhibitor (SSRI) treatment.
  Other Names: Abilify
  Arms: Medication Augmentation
Drug: Bupropion — Medication augmentation with Wellbutrin (bupropion), in participants who have not responded to SSRI treatment.
  Other Names: Wellbutrin
  Arms: Medication Augmentation
Behavioral: Problem Solving Therapy — Weekly specialized psychotherapy
  Arms: Problem Solving Therapy

SUMMARY:
The purpose of this study is to compare the effectiveness of two different augmentation strategies of antidepressant treatment for depressed older adults who have not responded to an adequate trial of antidepressant medication. The first augmentation strategy is Problem Solving Therapy (PST), a 12-week psychotherapy treatment that has been shown to be effective in depressed older adults. The second augmentation strategy is medication augmentation, which will begin with six weeks of aripiprazole, an atypical antipsychotic medication that has also been shown to be effective in depressed older adults who have failed a trial of antidepressant medication.

DETAILED DESCRIPTION:
Depression is common in older adults, and antidepressant medication is only effective in about 60% of patients seeking treatment. The purpose of this study is to compare the effectiveness of two different augmentation strategies of antidepressant treatment for depressed older adults who have not responded to an adequate trial of antidepressant medication. The first augmentation strategy is Problem Solving Therapy (PST), a 12-week psychotherapy treatment that has been shown to be effective in depressed older adults. The second augmentation strategy is medication augmentation, which will begin with six weeks of aripiprazole, an atypical antipsychotic medication that has also been shown to be effective in depressed older adults who have failed a trial of antidepressant medication. If patients have not remitted at the end of the 6 week aripiprazole trial, the aripiprazole will be stopped and they will be started on bupropion for the remaining 6 weeks of the study. Both aripiprazole augmentation and bupropion augmentation in depressed older adults have been approved by the FDA. No study has compared the effectiveness of PST and medication augmentation strategies for depressed older adults who are non-responders to an adequate trial of antidepressant medication in the current episode of their depression.

ELIGIBILITY:
Inclusion Criteria:

* Ages 50-90, inclusive
* Current diagnosis of major depressive disorder or dysthymia
* Treatment with either citalopram 30/mg or duloxetine 60 mg/day (6 weeks total, with at least three weeks of treatment at that dose)
* Hamilton Rating Scale for Depression (HRSD) >= 14
* Willing and able to complete NP testing
* Willing and able to complete medical exam, EKG, blood tests, and urine screen
* Willing and able to give consent

Exclusion Criteria:

* Meets criteria for psychotic depression
* MMSE score <24
* Bipolar disorder, psychotic disorder, or OCD
* History of alcohol or drug dependence (excluding nicotine) within past six months
* Suicide attempt within past six months or HRSD item 2 score > 2
* Diagnosis of probable Alzheimer's disease
* Diagnosis of probable vascular dementia
* Acute, severe, or unstable medical illness
* Patients in psychotherapy
* Diagnosis of Parkinson's Disease
* Blood glucose >200 and/or total cholesterol >250

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08 (Estimated); Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Psychiatric Rating Scale for Depression | 12 weeks
  The Hamilton Depression Rating Scale (HAM-D) is used as a way of determining a patient's level of depression before, during, and after treatment. The scoring is based on the first 17 list items. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2.

SECONDARY OUTCOMES:
Wechsler Abbreviated Scale of Intelligence (WASI) Matrix Reasoning Test | 1 Day
  IQ test designed to assess specific and overall cognitive capabilities and is individually administered

CONTACTS AND LOCATIONS:
Overall Officials: Bret Rutherford, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States